CLINICAL TRIAL: NCT00409019
Title: A Prospective, Randomized, Trial to Investigate the Effect of Continued Adefovir Versus Combination Regimens of Telbivudine Plus Adefovir, and Telbivudine Plus Tenofovir in Patients With Chronic Hepatitis B and Suboptimal Viral Suppression (PROACTIV Study)
Brief Title: Trial of Telbivudine Combination Therapy vs. Continued Adefovir Monotherapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study cancelled: Withdrawn before enrollment of any participants
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDT600AUS05
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Study cancelled: Withdrawn before enrollment of any participants
  Interventions: Drug: Telbivudine
- 2 (Experimental): Study cancelled: Withdrawn before enrollment of any participants
  Interventions: Drug: Adefovir
- 3 (Experimental): Study cancelled: Withdrawn before enrollment of any participants
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Telbivudine — Study cancelled: Withdrawn before enrollment of any participants
  Arms: 1
Drug: Adefovir
  Arms: 2
Drug: Tenofovir
  Arms: 3

SUMMARY:
The purpose of this study is to find out if taking a combination of telbivudine and adefovir or tenofovir and telbivudine can lower the amount of Hepatitis B virus in patients that have been taking adefovir alone for at least 5 months and have had less than optimal responses. The safety of taking telbivudine and adefovir together or tenofovir and telbivudine together will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Documented compensated chronic hepatitis B defined by clinical history compatible with chronic hepatitis B
* Patient is currently receiving Hepsera (adefovir dipivoxil) and has received treatment continuously for a minimum of 5 months prior to screening.

Other inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis C, hepatitis D or HIV
* Patient previously received nucleoside(tide) therapy other than adefovir
* Patient previously received an interferon-based treatment or an investigational agent for hepatitis B in the preceding 12 months

Other exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals